CLINICAL TRIAL: NCT00781378
Title: Efficacy and Safety Evaluation of Low Dosage of Recombinant Tissue Plasminogen Activator (rt-PA) in the Treatment of Pulmonary Thromboembolism: A Multi-Center, Randomized Controlled Trial in China
Brief Title: Low Dosage of rt-PA in the Treatment of Pulmonary Thromboembolism in China
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Chen WANG, Beijing Chao-Yang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2001BA703B13; 2004BA703B07
Record Dates: First submitted 2008-10-21; First posted 2008-10-29 (Estimated); Last update posted 2008-10-29 (Estimated); Status verified 2008-10

CONDITIONS: Pulmonary Embolism; Thromboembolism
Keywords: Thrombolytic therapy; Recombinant tissue plasminogen activator; Efficacy; Safety
MeSH Terms: conditions — Pulmonary Embolism; Thromboembolism | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Active Comparator): rt-PA 100 mg continuous intravenous infusion for 2 hours
  Interventions: Drug: rt-PA
- group 2 (Experimental): rt-PA 50 mg continuous intravenous infusion for 2 hours
  Interventions: Drug: rt-PA

INTERVENTIONS:
Drug: rt-PA — rt-PA 100 mg continuous intravenous infusion for 2 hours
  Other Names: Recombinant tissue plasminogen activator
  Arms: Group 1
Drug: rt-PA — rt-PA 50 mg continuous intravenous infusion for 2 hours
  Other Names: Recombinant tissue plasminogen activator
  Arms: group 2

SUMMARY:
Recombinant tissue plasminogen activator (rt-PA) is currently the most commonly used thrombolytic drug in patients with pulmonary thromboembolism (PTE). Optimal dosing with maximal benefits and minimal risks is of great importance. Considering the lower body weight in general Chinese population, we compared the efficacy and safety of lower dose rt-PA 50mg/2h regimen with the FDA-approved rt-PA 100mg/2h regimen in selected PTE patients.

DETAILED DESCRIPTION:
Pulmonary thromboembolism (PTE) is a severe and common clinical problem with substantial morbidity and mortality both in US and in Europe. Used to be considered as a rare disease in China, PTE has been increasingly diagnosed in recent years due to the increased awareness and the improvement of imaging techniques. PTE is life threatening without proper intervention at the early onset. Effective treatment can decrease the mortality and the complication of chronic thromboembolic pulmonary hypertension (CTEPH).

Recombinant tissue-type plasminogen activator (rt-PA) is currently the most commonly used drug for PTE thrombolysis. Like most thrombolytic medications, rt-PA carries a risk of significant bleeding, which is dose dependent. Thus, optimal dosing that can maximize benefits and minimize risks is of great importance. There is substantial controversy and debate regarding the optimal rt-PA dosage for thrombolytic therapy and whether the same dose should be used in all patients. Low dose of intravenous rt-PA for thrombolysis after acute myocardial infarction (AMI) had been suggested by previous studies. Experimental and clinical studies have indicated that a lower dose of rt-PA bolus may be potentially safer, and yet equally effective then the 2-h 100 mg rt-PA continuous infusion for PTE.

Considering lower body weight in Chinese population, a lower dose of 50mg rt-PA/2h may exhibit similar efficacy and safety as 100mg/2-h rt-PA for treating acute PTE in this population. We, therefore, compared these two regimens in a multi-center, randomized, controlled trial. The efficacy was assessed by the improvement of the right ventricular function on echocardiograms, perfusion defect score of lung V/Q scans or quantitative computed tomographic (CT) evaluation, safety was evaluated by incidence of major or minor bleeding, death rate, and PTE recurrence on 24h,14d after treatment.

110 patients will be randomized in the study. The patients included in the study will be randomized, in a double blind fashion, to receive rt-PA 100mg 2h (55 patients) or rt-PA50mg 2h(55 patients).Study treatment should be administered within 72 hours from echocardiography. Echocardiography will be repeated at 24 hours and 14 days from rt-PA injection. A Follow-up visit at 14 days from randomization will include: clinical history, physical examination and ECG and an echocardiographic examination CTPA and V/Q scan.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 75
* symptomatic PE confirmed by: a high probability ventilation-perfusion lung scanning (V/Q scan) or the presence of intraluminal filling defect on spiral computed tomographic pulmonary angiography (CTPA)
* PTE patients with haemodynamic instability, or cardiogenic shock
* anatomic obstruction more than 2 lobes on CTPA, or defect more than 7 segments on V/Q scan combined with evidence of right ventricular dysfunction(RVD) and pulmonary hypertension on echocardiography
* written informed consent

Exclusion Criteria:

* active bleeding or spontaneous intracranial hemorrhage
* major surgery, organ biopsy or recent puncture of a non-compressible vessel less than 10 days
* cerebral arterial thrombosis within 2 months
* gastro-intestinal bleeding within 10 days
* major trauma within the past 15 days
* neurosurgery or ophthalmologic operation with 30 days
* uncontrolled hypertension (systolic blood pressure > 180 mmHg and/or diastolic blood pressure > 110 mmHg)
* recent external cardiac resuscitation manoeuvres
* platelet count < 100 000/mm3 at admission
* pregnancy, puerperium or lactation with 2 weeks
* infectious pericarditis or endocarditis
* severe hepatic and kidney dysfunction
* hemorrhagic retinopathy due to diabetes
* a known bleeding disorder

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2002-06; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
The improvement of the right hart function on echocardiograms | within the 1st 14 days
Perfusion defect score of lung V/Q scans | within the 1st 14 days
Quantitative computed tomographic pulmonary angiography (CTPA) score on 2d, 14d after treatment. | within the 1st 14 days

SECONDARY OUTCOMES:
Major or minor bleeding | within 1st 14 days
PE recurrence | within the 1st 14 days
Death | within the 1st 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Chen WANG, Prof, Principal Investigator — Beijing Institute of Respiratory Medicine,Beijing Chao-Yang Hospital,Capital Medical University
Locations (23):
- China (23):
  - Beijing Chaoyang Hospital, Capital University of Medical Sciences, Beijing, Beijing Municipality
  - Beijing University People's Hospital, Beijing, Beijing Municipality
  - Peking Union Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - The Omni-hospital of Air-force, Beijing, Beijing Municipality
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Guangzhou Institute of Respiratory Disease, Guangdong, Guangzhou
  - The Second Affiliated Hospital of Hebei University, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Zhengzhou University:, Zhengzhou, Henan
  - Shenyang Military Hospital, Shenyang, Liaoning
  - The Affiliated Hospital of Shenyang Medical University, Shenyang, Liaoning
  - The Affiliated Hospital of Ningxia Medical University, Yinchuang, Ningxia
  - Shangdong Yantaishan Hospital, Yantai, Shandong
  - Qilu Hospital of Shandong University, Jinan, Shangdong
  - The First Affiliated Hospital of Jining Medical College, Jinan, Shangdong
  - The First Affiliated Hospital of Qingdao University CHENG Zhao-zhong, Qingdao, Shangdong
  - Shanghai Hospital of Lung Disease, Shanghai, Shanghai Municipality
  - Shanghai Ruijin Hospital HUANG Shao-guang, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Shanxi University, Taiyuan, Shanxi
  - The Second Affiliated Hospital of Shanxi University, Taiyuan, Shanxi
  - Tianjin Hospital of Medical Sciences, Tianjin, Tianjin Municipality
  - The Affiliated Hospital of Wenzhou Medical College, Wenzhou, Zhejiang
  - Zhejiang Shaoyifu Hospital, Hangzhou, Zhenjiang

REFERENCES:
- [Background] Pang BS, Wang C, Lu Y, Yang YH, Xing GH, Mao YL, Huang XX, Zhai ZG. [Changes of blood coagulative and fibrinolytic system and function of pulmonary vascular endothelium after therapy in patients with acute pulmonary thromboembolism]. Zhonghua Yi Xue Za Zhi. 2007 Nov 20;87(43):3074-8. Chinese. PMID 18261355
- [Background] Zhu L, Yang Y, Wu Y, Zhai Z, Wang C. Value of right ventricular dysfunction for prognosis in pulmonary embolism. Int J Cardiol. 2008 Jun 23;127(1):40-5. doi: 10.1016/j.ijcard.2007.06.093. Epub 2007 Aug 22. PMID 17716753
- [Background] Zhu L, Wang C, Yang Y, Wu Y, Zhai Z, Dai H, Pang B, Tong Z. Value of transthoracic echocardiography in therapy regimens evaluation in pulmonary embolism. J Thromb Thrombolysis. 2008 Dec;26(3):251-6. doi: 10.1007/s11239-007-0087-8. Epub 2007 Aug 21. PMID 17705052
- [Background] Zhu L, Yang YH, Wu YF, Zhai ZG, Wang C; National Project of the Diagnosis and Treatment Strategies for Pulmonary Thromboembolism investigators. Value of transthoracic echocardiography combined with cardiac troponin I in risk stratification in acute pulmonary thromboembolism. Chin Med J (Engl). 2007 Jan 5;120(1):17-21. PMID 17254482
- [Background] Zhai ZG, Wang C, Yang YH, Pang BS, Xiao B, Liu YM, Mao YL, Weng XZ. [Relationship between polymorphisms of plasminogen activator inhibitor-1 promoter gene and pulmonary thromboembolism in Chinese Han population]. Zhonghua Yi Xue Za Zhi. 2006 May 23;86(19):1313-7. Chinese. PMID 16796899
- [Background] Wang C, Cheng XS, Zhong NS. [Promoting the clinical and research work on pulmonary thromboembolism in China]. Zhonghua Jie He He Hu Xi Za Zhi. 2004 Nov;27(11):721-2. No abstract available. Chinese. PMID 15634378
- [Derived] Wang C, Zhai Z, Yang Y, Wu Q, Cheng Z, Liang L, Dai H, Huang K, Lu W, Zhang Z, Cheng X, Shen YH; China Venous Thromboembolism (VTE) Study Group. Efficacy and safety of low dose recombinant tissue-type plasminogen activator for the treatment of acute pulmonary thromboembolism: a randomized, multicenter, controlled trial. Chest. 2010 Feb;137(2):254-62. doi: 10.1378/chest.09-0765. Epub 2009 Sep 9. PMID 19741062